CLINICAL TRIAL: NCT01006551
Title: Ziprasidone in Early Onset Schizophrenia Spectrum Disorders
Acronym: ZEOSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Pfizer (Industry); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-0858; 2002-0012
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2009-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia Spectrum Disorders
MeSH Terms: conditions — Schizophrenia | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ziprasidone (Experimental)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — 20mg pills, dosing will be flexible, ranging from 10 to 160 mg divided BID or TID for the duration of the 52 week trial. In very rare cases, if the subject has shown some benefit and no side effects at a dose of 160mg and the treating clinician feels a further dose increase is necessary, the case would need to be presented to all of the other Principal Investigators for special consideration of further dose increases in 20 mg increments to an absolute maximal dose of 220mg.
  Other Names: Geodon

SUMMARY:
This is an open trial of ziprasidone (ZIP) in children and adolescents. It is designed to provide pilot data on the magnitude of ZIP's antipsychotic effects in psychotic youth, dosing ranges, acute safety, and tolerability. This would then inform the design of a rigorous, randomized controlled trial of ZIP in the pediatric population. The primary study hypothesis is that the proportion of pediatric subjects responding to treatment with ziprasidone will be comparable or greater than reported in trials of ziprasidone in adults.

DETAILED DESCRIPTION:
The study will consist of two phases: an eight week acute phase and a 44 week continuation phase for those subjects who show a response during the first eight weeks. All treatment will be open label and monitored by research clinicians with expertise in treating psychotic youth. The initial titration is relatively slow to minimize side effects. A flexible dose strategy in which each individual's ultimate dose is determined by his/her response and side effects will be used. The maximal dose will be 160mg split as a BID dose. We estimate that the average dose will be 120mg/d. Concurrent use of benztropine, propranolol, and benzodiazepines (lorazepam and clonazepam) will be permitted as needed to treat any emergent extrapyramidal side effects and agitation. Concurrent use of antidepressants and mood stabilizers will be permitted in those subjects who have been on stable doses of antidepressants or mood stabilizers for at least four weeks at time of entry, or those with emergence of significant affective symptoms during the maintenance phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Between 6 and 19 years old, male or female.
* Significant psychotic symptoms defined by a behavior score of at least 4 (moderate) on at least one of the psychotic items of Positive and Negative Symptom Scale (PANSS) at baseline.
* Subjects will meet DSM IV criteria for schizophrenia, schizoaffective disorder, or schizophreniform disorder.
* Subjects will be free of depot antipsychotic medication for at least six months.
* Good physical health.
* The subject gives informed assent for the study and his/her guardian is able and willing to give informed consent.
* Mood stabilizing treatment (i.e., antidepressant, lithium, carbamazepine, valproate) will be permitted during the first eight weeks of the study only if the patient has been treated with the mood stabilizer for at least 30 days. Dosages will remain stable for the first 8 weeks unless change or discontinuation is clinically indicated.

Exclusion Criteria:

* A primary diagnosis of substance abuse or dependence.
* Known endocrinological or neurological conditions, which confound the diagnosis or are a contraindication to treatment with antipsychotics.
* Subjects with a clear history of intolerance or nonresponsiveness to ziprasidone.
* Subjects at serious, short term risk for suicide.
* Subjects who are pregnant or who refuse to practice contraception during the study.
* Subjects with known cardiac conduction problems especially prior QTc prolongation, known genetic risk for QTc prolongation or who are being treated with other agents that prolong the QTc. These agents include the antiarrhythmic agents: dofetilide (Tikosyn), sotalol (Betapace), quinidine (Quinaglute), or Class 1A and III antiarrhythmics; the antipsychotics mesoridazine (Serentil), thioridazine (Mellaril), chlorpromazine (Thorazine), droperidol (Inapsine), pimozide (Orap); the anti-infectives: sparfloxacin (Zagam), gatifloxacin (Tequin), moxifloxacin (Avelox), pentamidine (Pentam); the anti-malarials halofantrine (Halfan), mefloquine (Lariam); and arsenic trioxide (Trisenox), levomethadyl acetate (Orlaam), dolasetron mesylate (Anzemet), probucol (Lorelco-an antilipemic), and tacrolimus (Prograf).
* Subjects with a diagnosis of a pervasive developmental disorder or an autism screening questionnaire score >15, must have clear hallucinations or delusions.
* Subjects will be excluded if they meet criteria for a current major depressive episode.

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2002-12; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be responder status, defined as a CGI improvement score of 1 or 2, plus a 20 % reduction in the baseline PANSS score at week 8. | 8 weeks

SECONDARY OUTCOMES:
A correlational analysis will be done to examine the potential relationship between dose and treatment response, and reduction in positive and negative symptoms. | 52 weeks
Subsequent analyses will examine the ZEOSS week 0 visit scores to assess for further improvement in symptoms and ability to sustain response/prevent relapse in subjects who responded to but could not tolerate the prior antipsychotic. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (4):
- United States (4):
  - Harvard University, Medford, Massachusetts
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - University of Washington, Seattle, Washington